CLINICAL TRIAL: NCT01128283
Title: Temporal Behavior of Coagulation Factors, Cytokines and Tissue Injury Markers in Sepsis
Brief Title: Indicators of Inflammation and Coagulation in Sepsis
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Gary Kinasewitz, Principal Investigator, University of Oklahoma
Other Study IDs: 09681
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Sepsis
Keywords: Sepsis; organ failure; cytokines; clotting factors
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sepsis: Patients with severe sepsis
- Non-infected: ICU patients without evidence of infection

SUMMARY:
We will collect blood samples from patients with the diagnosis of sepsis and other ICU patients. We will describe the course of different mediator levels and organ injury markers and follow their progression throughout the course of the study.

DETAILED DESCRIPTION:
After informed consent is obtained 5 cc of blood is collected on the day of admission and on days 0, 1, 3, and 7 thereafter. Plasma is collected and frozen for the subsequent measurement of biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ICU

Exclusion Criteria:

* No blood draws scheduled
* Hemoglobin level < 6,5 gm/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2002-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Death | 30 days
  Survival at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Gary T. Kinasewitz, MD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Medical Center, Oklahoma City, Oklahoma, United States